CLINICAL TRIAL: NCT00785694
Title: Recurrence of Bladder Cancer After Transurethral Resection With Hexvix
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Rejected ethics approval in UK and Holland
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: GE-196-001
Record Dates: First submitted 2008-11-04; First posted 2008-11-05 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — 5-aminolevulinic acid hexyl ester

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- B (Experimental): One instillation of mitomycin C after transurethral resection in white and blue fluorescence light with Hexvix.
  Interventions: Drug: hexaminolevulinate
- A (No Intervention): Multiple instillations of mitomycin C after transurethral resection in white light alone.

INTERVENTIONS:
Drug: hexaminolevulinate — Instillation of 50mL of 8mM Hexvix into the bladder through a catheter.
  Other Names: Hexvix
  Arms: B

SUMMARY:
This is a randomised, comparative, multicentre study to determine if the early recurrence rate of intermediate-risk bladder cancer is similar in subjects treated with multiple instillations of mitomycin C after resection conducted under white light cystoscopy (group A) and subjects treated with 1 instillation of mitomycin C after resection conducted under white light and blue light cystoscopy (group B).

ELIGIBILITY:
Inclusion Criteria:

* The subject is not of childbearing potential and signed informed consent.
* Subject with 1 or more primary bladder tumours, confirmed on an outpatient cystoscopy or subjects with 1 or more recurrent bladder tumours appearing within 12 months of removal of a previous bladder tumour, confirmed on an outpatient cystoscopy.

Exclusion Criteria:

* The subject was previously included in this study.
* The subject has a history/is suspected to have TaG3 or greater than or equal to T1 tumours or carcinoma in situ (CIS).
* The subject is suspected to have single primary or single recurrent TaG1 tumours when recurrence occurs more than 1 year after initial diagnosis or previous recurrence.
* The subject has known tumours in the prostatic urethra, distal urethra, or upper urinary tract.
* The subject has gross haematuria.
* The subject has a history of porphyria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-12; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Rate of bladder cancer recurrence | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul Antonini, Study Director — GE Healthcare
Locations (1):
- GE Healthcare Medical Diagnostics, Vélizy-Villacoublay, Morane Saulnier, France